CLINICAL TRIAL: NCT01109342
Title: Extended Follow-Up for Participants in VRC HIV-1 Recombinant Adenovirus-5 Vector Vaccine Studies in Uganda
Brief Title: Extended Follow-Up of Participants in Preventive HIV Vaccine Studies in Uganda
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: RV 283/WRAIR 1631; 11698 (Registry Identifier: DAIDS ES Registry Number); RV 283
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Prevention; Vaccine; Recombinant Adenovirus-5; HIV Preventative Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccine Recipients: Participants received HIV preventive vaccine VRC-HIV ADV014-00-VP in previous trials RV 156A/WRAIR 1078A or RV 172/WRAIR 1218.
- Placebo Recipients: Participants received a placebo vaccine in previous trials RV 156A/WRAIR 1078A or RV 172/WRAIR 1218.

SUMMARY:
Two previous studies of an HIV preventive vaccine, the STEP study and the Phambili study, were halted because people who received the vaccine were more likely to become infected with HIV. Why this vaccine failed is still being researched, but one reason may be related to the recombinant Adenovirus type 5 (rAd5) virus vector used in the vaccine. Two trials of another HIV preventive vaccine that used a rAd5 virus vector were conducted in Uganda. This study will obtain follow-up safety information on participants in those trials.

DETAILED DESCRIPTION:
Two previous trials of an HIV preventive vaccine, referred to as the MRK rAd5 vaccine, were halted because people receiving the vaccine were at greater risk of HIV infection. The MRK rAd5 vaccine delivered parts of HIV inside a recombinant Ad5 (rAd5) virus vector, which is a modified version of a common virus that does not usually cause serious disease. Analyses of these trials found that the increased risk of HIV infection was seen only in male participants who already had detectable antibodies to Adenovirus type 5 (Ad5).

A different HIV preventive vaccine developed by the Vaccine Research Center (VRC) at the U.S. National Institutes of Health (NIH) also uses a rAd5 virus vector. Although this vaccine, referred to as VRC Ad5, uses a rAd5 virus vector, it is structured and delivered differently than the MRK rAd5 vaccine. In two trials in Uganda it has shown no serious side effects. This study will perform safety follow-ups on participants in these two trials, RV 156A/WRAIR 1078A and RV 172/WRAIR 1218. Participants who received either the vaccine or the placebo will be recruited in order to compare health and HIV status.

Participants in this study will complete eight clinic visits over 1 year and 2 weeks. Four visits will be completed at baseline and after 4, 8, and 12 months. During these visits, participants will be checked for health changes and complete a blood draw. As part of the blood tests performed, participants will be tested for HIV. Every 2 weeks after the four visits mentioned (on Days 14, 134, 254, and 374), participants will return to the clinic to receive the results of their HIV tests. On all eight visits, participants will also receive HIV risk reduction counseling.

ELIGIBILITY:
Inclusion Criteria:

* Participated in either of the following studies: (1) RV 156A/WRAIR 1078A, or (2) RV 172/WRAIR 1218
* Able to provide informed consent

Exclusion Criteria:

* Incapacitating illness precluding clinic visits

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People who received either vaccine or placebo in two previous trials:
  1. RV 156A/WRAIR 1078A "A Phase I Clinical Trial To Evaluate The Safety And Immunogenicity Of A Multiclade HIV-1 Recombinant Adenovirus-5 Vector Vaccine, VRC-HIVADV014-00-VP Administered Alone Or Administered As A Boost To A Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA009-00-VP, In Uninfected Adult Volunteers In Uganda," or
  2. RV 172/WRAIR 1218 "A Phase I/II Clinical Trial To Evaluate The Safety And Immunogenicity Of A Multiclade HIV-1 DNA Plasmid Vaccine, VRCHIVDNA016-00-VP, Boosted By A Multiclade HIV-1 Recombinant Adenovirus-5 Vector Vaccine, VRC-HIVADV014-00-VP, In HIV Uninfected Adult Volunteers In East Africa." (NCT00123968)
Sampling Method: Non-Probability Sample
Dates: Start 2010-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Laboratory measures of safety, as defined in protocol | Measured at baseline and on Days 120, 240, and 360
Product-related adverse and serious adverse experiences | Measured over 1 year follow-up
HIV and rAdenovirus type 5 (rAd5) T-cell and antibody immune responses | Measured at baseline and on Days 120, 240, and 360
Risk behaviors | Measured at baseline and on Days 120, 240, and 360
HIV status | Measured on Days 14, 134, 154, and 374

CONTACTS AND LOCATIONS:
Locations (1):
- Makerere University Walter Reed Project (MUWRP), Kampala, Uganda

REFERENCES:
- [Background] Buchbinder SP, Mehrotra DV, Duerr A, Fitzgerald DW, Mogg R, Li D, Gilbert PB, Lama JR, Marmor M, Del Rio C, McElrath MJ, Casimiro DR, Gottesdiener KM, Chodakewitz JA, Corey L, Robertson MN; Step Study Protocol Team. Efficacy assessment of a cell-mediated immunity HIV-1 vaccine (the Step Study): a double-blind, randomised, placebo-controlled, test-of-concept trial. Lancet. 2008 Nov 29;372(9653):1881-1893. doi: 10.1016/S0140-6736(08)61591-3. Epub 2008 Nov 13. PMID 19012954
- [Background] McElrath MJ, De Rosa SC, Moodie Z, Dubey S, Kierstead L, Janes H, Defawe OD, Carter DK, Hural J, Akondy R, Buchbinder SP, Robertson MN, Mehrotra DV, Self SG, Corey L, Shiver JW, Casimiro DR; Step Study Protocol Team. HIV-1 vaccine-induced immunity in the test-of-concept Step Study: a case-cohort analysis. Lancet. 2008 Nov 29;372(9653):1894-1905. doi: 10.1016/S0140-6736(08)61592-5. Epub 2008 Nov 13. PMID 19012957
- [Background] Robb ML. Failure of the Merck HIV vaccine: an uncertain step forward. Lancet. 2008 Nov 29;372(9653):1857-1858. doi: 10.1016/S0140-6736(08)61593-7. Epub 2008 Nov 13. No abstract available. PMID 19012958
- See also: Click here for information on study RV 172/WRAIR 1218 (NCT00123968) — http://www.clinicaltrials.gov/ct2/show/NCT00123968?term=VRC-HIVADV014-00-VP&cntry1=AF%3AUG&phase=0&rank=1